CLINICAL TRIAL: NCT01483755
Title: Delayed Angioplasty Postconditioning in STEMI Patients
Brief Title: Delayed Postconditioning
Acronym: PRIME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008.536/37
Record Dates: First submitted 2011-11-30; First posted 2011-12-01 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Myocardial Reperfusion Injury
Keywords: Myocardial infarction; Postconditioning
MeSH Terms: conditions — Myocardial Reperfusion Injury; Myocardial Infarction | interventions — Ischemic Postconditioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Postconditionned (Experimental): 36 postconditionned patients
  Interventions: Procedure: Postconditioning
- Conventional intervention (Sham Comparator): 36 control patients with conventional primary percutaneaous intervention (PCI)
  Interventions: Procedure: Percutaneaous intervention

INTERVENTIONS:
Procedure: Postconditioning — Postconditioning consists of four cycles of one minute balloon inflation followed by one minute of balloon deflation, with the initial inflation being started within the first minute after reopening of the culprit coronary artery.
  Arms: Postconditionned
Procedure: Percutaneaous intervention — Conventional primary percutaneaous intervention
  Arms: Conventional intervention

SUMMARY:
The investigators previously reported that angioplasty postconditioning reduces infarct size (cardiac enzyme release) in STEMI patients with a fully occluded coronary artery at hospital admission. Animal studies have suggested that the time window for applying brief episodes of ischemia and reperfusion aimed at triggering postconditioning's protection is very narrow, i.e. does not expand beyond 1 minute after reflow. We sought to address whether this window might be larger in humans, i.e. whether STEMI patients might be protected several minutes after undergoing spontaneous reperfusion before admission coronary angiography.

Therefore, STEMI patients (onset of chest pain less than 12 hours) with a TIMI flow grade > 1 were eligible for that study. Angioplasty postconditioning was completed as already published and infarct size was assessed by measuring cardiac enzymes release.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years old
* Male or female
* Presenting first myocardial infarction, with the beginning of pains < 12 hours,
* Requiring a revascularisation by primary angioplasty or " rescue " (after failure of thrombolysis) on LAD or RCA (not Circumflex coronary artery).
* TIMI flow grade at admission of 2 or 3
* LV angiography (RAO30°) before angioplasty.

Exclusion Criteria:

* Cardiac arrest before the angioplasty
* Cardiogenic shock
* Occlusion of the artery circumflex responsible for the infarction
* Visible collaterals to the area at risk
* Magnetic resonance imaging: contra indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Size of the infarct | Day 5 post reperfusion
  Size of the infarct estimated by magnetic resonance imaging at day 5 post-reperfusion

SECONDARY OUTCOMES:
Contractile functional recovery | 6 months after reperfusion
  Contractile functional recovery estimated by echocardiography at 6th month versus before discharge.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Service de Cardiologie, CHU d'Angers, Angers
  - Service d'explorations Fonctionnelles Cardiovasculaires, Hôpital Cardiologique Louis Pradel, Bron
  - Service de Cardiologie, Hôpital Arnaud de Villeneuve, Montpellier
  - Service de Cardiologie, Hôpital Emile Müller, Mulhouse
  - Service de Cardiologie, Hôpital Rangueil, Toulouse

REFERENCES:
- [Result] Roubille F, Mewton N, Elbaz M, Roth O, Prunier F, Cung TT, Piot C, Roncalli J, Rioufol G, Bonnefoy-Cudraz E, Wiedemann JY, Furber A, Jacquemin L, Willoteaux S, Abi-Khallil W, Sanchez I, Finet G, Sibellas F, Ranc S, Boussaha I, Croisille P, Ovize M. No post-conditioning in the human heart with thrombolysis in myocardial infarction flow 2-3 on admission. Eur Heart J. 2014 Jul 1;35(25):1675-82. doi: 10.1093/eurheartj/ehu054. Epub 2014 Feb 28. PMID 24585265